CLINICAL TRIAL: NCT02673671
Title: Measurement Of GI Myoelectric Activity In Patients At Risk For Or Who Have A Post-Operative Ileus (POI) - Monitoring/ Recording GI Myoelectric Activity For Early Detection of A POI
Brief Title: G-Tech Feasibility Study for Early Detection of a Post-op Ileus
Acronym: GTECHPOI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: G-Tech Corporation (Industry)
Collaborators: Eminence Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-2014-001
Record Dates: First submitted 2016-01-27; First posted 2016-02-04 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Post-operative Ileus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with unknown POI status consented pre-surgery: Up to 100 subjects may be consented prior to surgery who are planned to undergo gastrointestinal surgery or a planned surgery that does not involve the abdominal cavity. The investigator does not change the routine medical care of study participants.
  Interventions: Device: G-Tech Myoelectric recording device
- Subjects with known/unknown POI status consented post-surgery: Up to 50 subjects who have undergone gastrointestinal surgery or surgery not involving the abdominal cavity may be consented post- operatively during their hospital stay for this study.The investigator does not change the routine medical care of study participants.
  Interventions: Device: G-Tech Myoelectric recording device

INTERVENTIONS:
Device: G-Tech Myoelectric recording device — A minimum of three patches are placed on the abdomen of the patient to record myoelectric activity.
  Other Names: Gastro-intestinal electrical recording

SUMMARY:
This feasibility study is for the purpose of determining if the G-Tech Device can differentiate between normal return of GI activity post-operatively and the myoelectric activity in patients who develop a POI.

DETAILED DESCRIPTION:
While preventing the development of a POI is most important, POIs still occur; therefore, it is important to definitively diagnose a POI as early as possible during the post-operative course for treatment to prevent patient discomfort, complications, and extended hospital stay. The purpose of the G-Tech study is to determine if the G-Tech Device can detect a difference in the myoelectric signals from patients who develop a POI compared to those patients who do not develop a POI. It is anticipated that up to 20% of patients enrolled in this study and consented preoperatively, excluding screen failures, will show evidence of a post-operative ileus as detected by the G-Tech GutCheck Device and differentiate the myoelectric signals from the patients who do not develop a POI. Patients who are known to have developed a POI may also be selected for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent;
2. Eighteen (18) years of age or older;
3. Subject is willing and able to follow all study requirements;
4. Subject who will undergo or has undergone open or laparoscopic gastrointestinal surgery or surgery not involving the abdominal cavity.

Exclusion Criteria:

1. Subject is pregnant or suspects pregnancy;
2. Known allergy to medical grade adhesive;
3. Weight > 350 lbs (159 Kg);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include candidates who undergo GI surgery or other surgery outside not involving the abdominal cavity, who agree to the application of the G-Tech Device to be placed on his/her abdomen and meet all eligibility criteria as defined. Up to 100 subjects may be consented prior to surgery who are planned to undergo gastrointestinal surgery or a planned surgery that does not involve the abdominal cavity or following. Up to 50 subjects who have undergone gastrointestinal surgery or surgery not involving the abdominal cavity may be consented post-operatively during their hospital stay for this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-02; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Myoelectric activity pattern in POI patients versus non-POI patients | Up to 6 Days
  The resumption of motor activity in the stomach, small intestine, and colon post-operatively. The measurement is myoelectric signals measured at the skin surface similar to ECG recordings for the heart

SECONDARY OUTCOMES:
Anticipated Adverse Events | Up to 6 days
  Device related anticipated adverse events; such as, skin irritation due to adhesive from the skin patch.
UADEs | Up to 6 Days
  Unanticipated adverse device effects
Device Success | Up to 6 Days
  Device success defined as the ability to record GI myoelectric activity following GI surgery.

CONTACTS AND LOCATIONS:
Overall Officials: George Triadafilopoulos, MD, Principal Investigator — El Camino GI Medical Associates
Locations (1):
- El Camino Hospital, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No
Analyses planned to be presented at scientific meetings and published in peer reviewed medical journals.

REFERENCES:
- [Background] Bederman SS, Betsy M, Winiarsky R, Seldes RM, Sharrock NE, Sculco TP. Postoperative ileus in the lower extremity arthroplasty patient. J Arthroplasty. 2001 Dec;16(8):1066-70. doi: 10.1054/arth.2001.27675. PMID 11740765
- [Background] Doorly MG, Senagore AJ. Pathogenesis and clinical and economic consequences of postoperative ileus. Surg Clin North Am. 2012 Apr;92(2):259-72, viii. doi: 10.1016/j.suc.2012.01.010. PMID 22414412
- [Background] Behm B, Stollman N. Postoperative ileus: etiologies and interventions. Clin Gastroenterol Hepatol. 2003 Mar;1(2):71-80. doi: 10.1053/cgh.2003.50012. PMID 15017498
- [Background] Frantzides CT, Cowles V, Salaymeh B, Tekin E, Condon RE. Morphine effects on human colonic myoelectric activity in the postoperative period. Am J Surg. 1992 Jan;163(1):144-8; discussion 148-9. doi: 10.1016/0002-9610(92)90267-u. PMID 1733363
- [Background] Tropskaya NS and Popova TS. (2012). Postoperative Ileus: Pathophysiology and Treatment in Current Concepts in Colonic Disorders, Dr. Godfrey Lule (Ed.), ISBN: 978-953-307-957-8, InTech, Available from: http://www.intechopen.com/books/current-concepts-in-colonic-disorders/postoperative-ileus-pathophysiologyand-treatment.
- [Background] Waldhausen JH, Shaffrey ME, Skenderis BS 2nd, Jones RS, Schirmer BD. Gastrointestinal myoelectric and clinical patterns of recovery after laparotomy. Ann Surg. 1990 Jun;211(6):777-84; discussion 785. doi: 10.1097/00000658-199006000-00018. PMID 2357140